CLINICAL TRIAL: NCT01468792
Title: Hemodynamic Changes in Connective Tissue Disease
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 23-409 ex 10/11; 23-409 ex 10/11 (Other Grant/Funding Number: MUG)
Record Dates: First submitted 2011-11-07; First posted 2011-11-09 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Systemic Sclerosis
Keywords: systemic sclerosis; pulmonary arterial hypertension
MeSH Terms: conditions — Scleroderma, Systemic; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study serves the identification of early forms of pulmonary arterial hypertension (PAH) in connective tissue disease and the hemodynamic follow-up of the investigated patients. The basic hypothesis is that PAH may start with a remodeling of small pulmonary arteries, which leads to a stiffening of the vessels, indicated by the inability to vasodilatation and thus a disproportional increase in pulmonary pressure during exercise. Recent studies have shown that a proportion of such patients may develop manifest PAH within a few years. The early identification of these patients and the understanding of the natural course of the disease may improve prognosis. The aim of the present study is to investigate hemodynamic and clinical changes in patients with connective tissue disease in a time interval of 3-5 years with a focus on the development of pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Patients with systemic sclerosis, mixed connective tissue disease, (systemic lupus erythematodes) SLE or overlap syndrome
* Existing exercise Doppler echocardiography or/and right heart catheterization 3-5 years before inclusion

Exclusion Criteria:

* - Severe lung or bronchial disease (FEV1 <60%)
* Systolic LV dysfunction (LVEF <50%) or diastolic dysfunction > grade I
* Valvular defect > grade I (except for tricuspid- or pulmonary insufficiency)
* Uncontrolled systemic arterial hypertension (at rest >150 mmHg systolic or 95 mmHg diastolic)
* Uncontrolled ventricular arrhythmias
* Uncontrolled bradycardia or tachycardia supraventricular arrhythmias
* Myocardial infarction within the last 12 months
* Pulmonary embolism within the last 12 months
* Relevant changes in hemodynamic therapy or major surgery within the last 12 weeks
* Musculoskeletal or peripheral vessel disorders which complicates an ergometry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with known systemic sclerosis and without known pulmonary hypertension
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2011-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
systolic pulmonary pressure at 50 W | 3-5 years
  change of systolic pulmonary arterial pressure after 3-5 years

SECONDARY OUTCOMES:
peak (oxygen uptake) VO2 | 3-5 years
  change of peak VO2 after 3-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz / Pulmonology, Graz, Austria

REFERENCES:
- [Derived] Kovacs G, Avian A, Wutte N, Hafner F, Moazedi-Furst F, Kielhauser S, Aberer E, Brodmann M, Graninger W, Foris V, Olschewski A, Olschewski H. Changes in pulmonary exercise haemodynamics in scleroderma: a 4-year prospective study. Eur Respir J. 2017 Jul 13;50(1):1601708. doi: 10.1183/13993003.01708-2016. Print 2017 Jul. PMID 28705939